CLINICAL TRIAL: NCT05230849
Title: Effectiveness of a Treatment Plan of Neurological Physiotherapy in Conjunction With Ultrasound-guided Dry Needling in Stroke Patients.
Brief Title: Effectiveness of a Treatment Plan of Neurological Physiotherapy in Conjunction With Ultrasound-guided Ultrasound-guided Dry Needling in Stroke Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica de Ávila (Other)
Responsible Party: Principal Investigator, JORGE VELAZQUEZ SAORNIL, Principal Investigator, Universidad Católica de Ávila
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13/01/2022
Record Dates: First submitted 2022-01-13; First posted 2022-02-09 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Neurological Disorder
Keywords: dry needling; physiotherapy techniques; anterior tibial muscle; posterior tibial muscle; Neurological Disorder
MeSH Terms: conditions — Nervous System Diseases | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Simple blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Active Comparator): conventional physiotherapy treatment
  Interventions: Other: convencional treatment
- dry needling treatment (Experimental): group that includes a dry needling treatment on the tibialis anterior and posterior muscles.
  Interventions: Device: dry needling

INTERVENTIONS:
Device: dry needling — is a physiotherapy treatment for neurological patients and studies the efficacy of dry needling by studying several pre-treatment and post-treatment variables after the experimental treatment.
  Arms: dry needling treatment
Other: convencional treatment — is a physiotherapy treatment for neurological patients
  Arms: control group

SUMMARY:
The aim of the study is to assess the efficacy of dry needling in stroke patients in combination with intensive neurological physiotherapy.

together with intensive neurological physiotherapy treatment. Randomised and blinded experimental study control group where the sample recruited was 20 patients, who were randomly assigned to a control group.

randomly assigned to a control group, where they received intensive treatment, or to an intervention group, where they received intervention group, where they received ultrasound-guided dry needling of the tibialis anterior and posterior muscles followed by an intensive followed by intensive neurological physiotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* left middle cerebral artery infarction
* impaired stability during walking
* patient between the age range 18 to 70 years old

Exclusion Criteria:

* patient under 18 years of age
* patients over 70 years of age
* undiagnosed left middle cerebral artery infarction patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-02-12 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
walking motor skills | 1 hour
  measures of gait motor ability using the time up ang go test.
spasticity | 1 hour
  measurements of spatiality using the modified Ashworth scale

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica de Ávila, Ávila, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edmiaston J, Connor LT, Steger-May K, Ford AL. A simple bedside stroke dysphagia screen, validated against videofluoroscopy, detects dysphagia and aspiration with high sensitivity. J Stroke Cerebrovasc Dis. 2014 Apr;23(4):712-6. doi: 10.1016/j.jstrokecerebrovasdis.2013.06.030. Epub 2013 Jul 30. PMID 23910514
- [Background] Hernandez-Ortiz AR, Ponce-Luceno R, Saez-Sanchez C, Garcia-Sanchez O, Fernandez-de-Las-Penas C, de-la-Llave-Rincon AI. Changes in Muscle Tone, Function, and Pain in the Chronic Hemiparetic Shoulder after Dry Needling Within or Outside Trigger Points in Stroke Patients: A Crossover Randomized Clinical Trial. Pain Med. 2020 Nov 1;21(11):2939-2947. doi: 10.1093/pm/pnaa132. PMID 32488238
- [Result] Sanchez-Mila Z, Salom-Moreno J, Fernandez-de-Las-Penas C. Effects of dry needling on post-stroke spasticity, motor function and stability limits: a randomised clinical trial. Acupunct Med. 2018 Dec;36(6):358-366. doi: 10.1136/acupmed-2017-011568. Epub 2018 Jul 9. PMID 29986902
- [Result] Cuenca Zaldivar JN, Calvo S, Bravo-Esteban E, Oliva Ruiz P, Santi-Cano MJ, Herrero P. Effectiveness of dry needling for upper extremity spasticity, quality of life and function in subacute phase stroke patients. Acupunct Med. 2021 Aug;39(4):299-308. doi: 10.1177/0964528420947426. Epub 2020 Aug 20. PMID 32815384
- [Result] Mendigutia-Gomez A, Martin-Hernandez C, Salom-Moreno J, Fernandez-de-Las-Penas C. Effect of Dry Needling on Spasticity, Shoulder Range of Motion, and Pressure Pain Sensitivity in Patients With Stroke: A Crossover Study. J Manipulative Physiol Ther. 2016 Jun;39(5):348-358. doi: 10.1016/j.jmpt.2016.04.006. Epub 2016 May 7. PMID 27167369
- [Result] Salom-Moreno J, Sanchez-Mila Z, Ortega-Santiago R, Palacios-Cena M, Truyol-Dominguez S, Fernandez-de-las-Penas C. Changes in spasticity, widespread pressure pain sensitivity, and baropodometry after the application of dry needling in patients who have had a stroke: a randomized controlled trial. J Manipulative Physiol Ther. 2014 Oct;37(8):569-79. doi: 10.1016/j.jmpt.2014.06.003. Epub 2014 Sep 8. PMID 25199825
- [Result] Fakhari Z, Ansari NN, Naghdi S, Mansouri K, Radinmehr H. A single group, pretest-posttest clinical trial for the effects of dry needling on wrist flexors spasticity after stroke. NeuroRehabilitation. 2017;40(3):325-336. doi: 10.3233/NRE-161420. PMID 28222554
- [Result] Wu WX, Zhou CY, Wang ZW, Chen GQ, Chen XL, Jin HM, He DR. Effect of Early and Intensive Rehabilitation after Ischemic Stroke on Functional Recovery of the Lower Limbs: A Pilot, Randomized Trial. J Stroke Cerebrovasc Dis. 2020 May;29(5):104649. doi: 10.1016/j.jstrokecerebrovasdis.2020.104649. Epub 2020 Feb 27. PMID 32115341
- [Result] Lee P, Tse CY. Calibration of wrist-worn ActiWatch 2 and ActiGraph wGT3X for assessment of physical activity in young adults. Gait Posture. 2019 Feb;68:141-149. doi: 10.1016/j.gaitpost.2018.11.023. Epub 2018 Nov 19. PMID 30476691
- [Derived] Sanchez Mila Z, Velazquez Saornil J, Campon Chekroun A, Barragan Casas JM, Frutos Llanes R, Castrillo Calvillo A, Lopez Pascua C, Rodriguez Sanz D. Effect of Dry Needling Treatment on Tibial Musculature in Combination with Neurorehabilitation Treatment in Stroke Patients: Randomized Clinical Study. Int J Environ Res Public Health. 2022 Sep 28;19(19):12302. doi: 10.3390/ijerph191912302. PMID 36231604